CLINICAL TRIAL: NCT03834675
Title: Are Peripherally Inserted Central Catheters (PICC) Suitable for Cardiac Output Assessment With Trans-pulmonary Thermodilution
Brief Title: Suitability of PICC for Transpulmonary Thermodilution Compared to CICC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Claudio Sandroni (Unknown); Sofia Cacciola (Unknown); Antonio Maria Dell Anna (Unknown); Mauro Pittiruti (Unknown); Maria Giuseppina Annetta (Unknown); Cesare Colosimo (Unknown); Massimo Antonelli (Unknown)
Responsible Party: Principal Investigator, Dr.ssa Sonia D'Arrigo, Medical Doctor - PhD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: PICC -CICC for TPTD
Record Dates: First submitted 2019-02-05; First posted 2019-02-08 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2019-02

CONDITIONS: Peripherally Inserted Central Catheters; CVC; Transpulmonary Thermodilution; Hemodynamic Monitoring
Keywords: PICC; shock; cardiac output
MeSH Terms: conditions — Shock

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: transpulmonary thermodilution — Thermodilution was attempted via PICC and via CICC

SUMMARY:
Peripherally inserted central catheters (PICCs) are increasingly used in intensive care unit (ICU) as an alternative to centrally inserted central catheters (CICCs) for intravenous infusion. In the present study we try to assess their reliability for measuring cardiac index (CI) with trans-pulmonary thermodilution (TPTD) technique.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (≥18 years) admitted to the ICU
* Patients requiring hemodynamic monitoring using EV1000TM
* Patients having both PICC and CICC in place (these patients had their PICC replaced with a CICC, usually at the time of ICU admission, or vice versa, usually at the end of their ICU stay, and were enrolled immediately after the placement of the new device before the previous one was removed)

Exclusion Criteria:

* body weight <40 kg
* severe aortic regurgitation or intra-cardiac shunt
* treatment with an intra-aortic balloon pump
* contraindication for placement of PICC, CICC or a femoral arterial catheter
* abdominal aneurism
* extracorporeal circulation
* pregnancy
* lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Cardiac Index comparison via PICC | One hour
  comparison of hemodynamic measurements made by the TPTD from the VolumeView/EV1000TM system via PICC vs. CICC.

SECONDARY OUTCOMES:
Comparison 4Fr PICCs to CICC | one hour
  Comparison of single-lumen 4 Fr PICCs to CICC in their reliability of assessing cardiac output
Comparison 5Fr PICCs to CICC | one hour
  Comparison of dual-lumen 5 Fr PICCs to CICC in their reliability of assessing cardiac output

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Antonelli, MD, Study Chair — Università Cattolica del sacro Cuore- Fondazione Policlinico Universitario A. Gemelli IRCSS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] D'Arrigo S, Sandroni C, Cacciola S, Dell'Anna AM, Pittiruti M, Annetta MG, Colosimo C, Antonelli M. Are Peripherally Inserted Central Catheters Suitable for Cardiac Output Assessment With Transpulmonary Thermodilution? Crit Care Med. 2019 Oct;47(10):1356-1361. doi: 10.1097/CCM.0000000000003917. PMID 31356470